CLINICAL TRIAL: NCT01112124
Title: Behaviors of Children Ages 15 Months to Five Years Around Microwave Ovens
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 14594B
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Scald Burn Injuries
Keywords: Typical; Development; Microwave; Children; Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the typical behavior of children ages 15 months to five years around a microwave oven. The UCH Burn and Complex Wound Center has observed scald burn injuries in young children operating and/or removing hot liquids from microwave ovens. The knowledge we hope to gain is the developmental age that a child is able to open and/or operate a microwave oven safely. This work may influence future microwave oven design to protect young children from microwave-related scald burn injuries. These injuries have resulted in visits to the emergency room, stays in the hospital and debridement and skin grafting procedures in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* a microwave oven in the child's home environment,
* age appropriate development,
* intact visual acuity, and
* English speaking.

Exclusion Criteria:

* developmental delay,
* non-English speaking.

Ages: 15 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Typically developing children ages 15 months to 5 years born full term
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Gottlieb, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States